CLINICAL TRIAL: NCT05561985
Title: Expanded Access Use of Itacitinib to Treat a Single Patient With STAT1 Gain of Function (GOF) Disease
Status: Available | Type: Expanded Access
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: I-39110-19-03
Record Dates: First submitted 2022-09-22; First posted 2022-09-30 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: STAT1 Gain-of-Function Disease
Keywords: STAT1 GOF disease
MeSH Terms: interventions — itacitinib; INCB039110

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Itacitinib
  Other Names: INCB039110

SUMMARY:
Expanded access use of Itacitinib to treat a single patient with aplastic anemia.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Forbes Satter, MD, Principal Investigator — Baylor College of Medicine - Texas Children's Hospital